CLINICAL TRIAL: NCT04722965
Title: Randomized Clinical Trial for the Treatment of Lower Transsphincteric Perianal Fistula Using Fistulotomy With Marsupialization vs Open Wound
Brief Title: Treatment of Lower Transsphincteric Perianal Fistula: Fistulotomy With Marsupialization vs Open Wound
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Feasibility problems to patients recruitment.
Sponsor: Consorci Sanitari de l'Alt Penedès i Garraf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CSAPG-13
Record Dates: First submitted 2021-01-21; First posted 2021-01-25 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Perianal Fistula; Transsphincteric Anal Fistula
Keywords: low transsphincteric anal fistula; fistulotomy; marsupialization; perianal fistula

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fistulotomy with marsupialization (Active Comparator): 40 patients with a simple low transsphincteric anal fistula. A fistulotomy with marsupialization is performed.
  Interventions: Procedure: Fistulotomy with marsupialization
- Fistulotomy with open wound (Active Comparator): 40 patients with a simple low transsphincteric anal fistula. A fistulotomy leaving the wound open is performed.
  Interventions: Procedure: Fistulotomy with open wound

INTERVENTIONS:
Procedure: Fistulotomy with marsupialization — A probe is placed in the fistula tract and it's laid open over that probe. The tract is curretted. Wound edges are sutured to the bottom of the fistula using interrupted sutures of vicryl 3-0 completing the marsupialization.
  Arms: Fistulotomy with marsupialization
Procedure: Fistulotomy with open wound — A probe is placed in the fistula tract and it's laid open over that probe. The tract is curretted. The wound is left open.
  Arms: Fistulotomy with open wound

SUMMARY:
This study will compare the results of marsupialization versus open wound after fistulotomy in low transsphincteric perianal fistulas.

DETAILED DESCRIPTION:
This is a multi-center triple blinded randomized clinical trial in which we'll compare two techniques for the treatment of simple low transsphincteric perianal fistulas. 40 patients will undergo a fistulotomy with marsupialization and 40 patients will undergo a fistulotomy with open wound. There will be an inclussion visit in which personal information will be recorded and the consent will be signed. Randomization will be done after inclusion, following a balanced blocks model. Information of the surgery technic won't be available for the investigator. The patients will have a journal in which they'll write their postoperative symptoms. Follow up will be done at weeks 2, 4 and 6 by the main investigator of each center. Data will be based in clinical examination, patient's diary and medical records. Statistical analysis of the primary outcome will be based in a superiority analysis using the Mantel-Cox test, or in case needed, a multivariate Cox regression analysis. The secondary outcomes will be analyzed by comparing times, percentages, mean or median with parametric or non parametric tests as it corresponds.

ELIGIBILITY:
Inclusion Criteria:

* Low transsphinteric perianal fistula, defined as a single tract in the lower third of the anal sphincter, confirmed by ultrasound and intraoperative evaluation.
* Ability to understand the study, to sign the consent and to complete the follow-up.

Exclusion Criteria:

* Under 18 years of age.
* Complex/recurrent fistula.
* Patients in which by clinical criteria is decided not to perform a fistulotomy.
* Anorectal malignancy.
* Crohn's desease.
* ASA IV or other contraindication for surgery.
* Inmunosuppressed patients or in treatment with steroids or cytotoxic drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Wound healing time | 6 weeks
  Comparisson of the time it takes for the wound to not have areas without epithelium after the fistulotomy between the group with marsupialization and the open wound group.

SECONDARY OUTCOMES:
Postoperative pain | 6 weeks
  Maximum pain experienced by the patient in the postoperative period measured by the visual scale of pain.
Return to daily activities | 6 weeks
  Days it takes the patients to return their daily activities (e.g. job).
Operating time | 60 minutes
  Time the surgery takes since the assessment of the fistula tract to the beginning of dressing of the postoperative wound. It's measured in minutes.
Hospitalization time | 2 days
  Days the patient has to stay admitted in the hospital.
Bleeding of the postoperative wound | 6 weeks
  Number of bleeding episodes that require more changing of the dressings or assistance of a medical professional.
Anal incontinence | 6 weeks
  Postoperative anal incontinence measured by the Browning and Parks incontinence scale: I: normal continence, II: Continent for solid and liquid stools but not for flatus, III: Continent for solid stools only, IV: Complete incontinence.
Frequency of dressing change | 6 weeks
  Number of times per day a patient needs a dressing change
Who performs the dressing change | 6 weeks
  Indicate who performs the dressing change: Patient, family member or medical professional.
Postoperative wound infection | 6 weeks
  Presence of erythema, induration surrounding the wound or suppuration with or without an isolated pathogenic microorganism.
Recurrence of the fistula | 1 year
  Reappearance of the fistula after complete healing of the surgical wound within the period of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Gonzales, MD, Principal Investigator — CSAPG
Locations (1):
- Consorci Sanitari Alt Penedes i Garraf, Sant Pere de Ribes, Barcelona, Spain